CLINICAL TRIAL: NCT04452916
Title: Physiological Response to Prolonged Fasting in Healthy Volunteers
Brief Title: Physiological Response to 5 Days Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sylvia Bähring, PhD, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LEANER
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Waiting list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Active Comparator): Starts immediately with 5 days of Buchinger fasting
  Interventions: Other: Buchinger fasting
- Waiting list control (Placebo Comparator): Starts with 5 days of Buchinger fasting after a waiting period of 12 weeks
  Interventions: Other: Buchinger fasting

INTERVENTIONS:
Other: Buchinger fasting — Caloric intake of < 250 kcal/d for 5 days

SUMMARY:
To investigate energy metabolism, anthropometry, blood pressure, gut microbiome, serum metabolome, glucose variability and neural mechanisms of food choice and mood before and after 5 days of fasting as well as their persistence in healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 20-50 years
* Body mass index 20-30 kg/m2

Exclusion Criteria:

* Clinically relevant heart, lung, liver, and kidney diseases
* Any prescribed medication (except for oral contraceptives)
* Current or chronic infection
* Intake of antibiotics within 6 months before study entry
* Fasting week within 6 months before study entry
* Habitual use of dietary supplements
* Food intolerances
* Pregnancy, lactation
* Vegan diet
* Smokers
* In addition for fMRI: sensorineural hearing loss, tinnitus, metal implants, electric devices

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure | 6-th day of fasting compared to baseline
  Measured by indirect calorimetry (kcal/d)

SECONDARY OUTCOMES:
Resting Energy Expenditure - Recovery | 12 weeks after fasting compared to baseline
  Measured by indirect calorimetry (kcal/d)
Resting Respiratory Exchange Ratio | 6-th day of fasting and 28 days after fasting compared to baseline
  Measured by indirect calorimetry
Office systolic blood pressure | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Mean of five consecutive blood pressure measurements (mmHg)
Office diastolic blood pressure | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Mean of five consecutive blood pressure measurements (mmHg)
Fecal microbiome composition | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Measured by 16S Sequencing
Fecal and serum metabolome | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Measured by mass spectrometry
Change in immune cell phenotypes | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Peripheral blood effector T cell frequencies (Percent)
Glucose variability | From 3 days before until 6 days after fasting
  Measured by continuous glucose monitoring over 14 days
Neural correlates of emotion processing | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Measured by functional Magnetic Resonance Imaging
Neural correlates of food-specific delay discounting | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Measured by functional Magnetic Resonance Imaging
Perceived Stress Questionaire (PSQ) | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Range 0-100, with 0 indicating no perceived stress
Perceived Self Efficiency | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Range 10-40, with 40 indicating highest self efficiency
PANAS Positive Affect Subscale (GESIS Panel) | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Range 10-50, with 50 indicating highest positive affect
PANAS Negative Affect Subscale (GESIS Panel) | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Range 10-50, with 50 indicating highest negative affect
International Physical Activity Questionaire (IPAQ, long version) | 6-th day of fasting and 12 weeks after fasting compared to baseline
  Time for moderate and vigorous activity (hours, minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Bähring, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.